CLINICAL TRIAL: NCT07080697
Title: The Impact of Splenectomy on Debridement Efficacy, Perioperative Recovery, and Prognosis in Patients With Acute Necrotizing Pancreatitis Complicated by Pancreatic Sinistral Portal Hypertension
Brief Title: A Study to Evaluate Splenectomy on Debridement for Acute Necrotizing Pancreatitis With Pancreatic Sinistral Portal Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Director physician, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT20250028C
Record Dates: First submitted 2025-07-04; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Acute Necrotizing Pancreatitis; Portal Hypertension
Keywords: Acute Necrotizing Pancreatitis; Pancreatic Sinistral Portal Hypertension; Debridement; Splenectomy
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing; Hypertension, Portal | interventions — Splenectomy

STUDY DESIGN:
Intervention Model Description: One group will receive open debridement combined with distal pancreatectomy and total splenectomy, the other group will receive open debridement alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Splenectomy group (Experimental): Open Debridement combined with Distal Pancreatectomy and Total Splenectomy
  Interventions: Procedure: Splenectomy
- Control group (Experimental): Open Debridement alone
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Splenectomy — Open Debridement combined with distal pancreatectomy and total splenectomy
  Arms: Splenectomy group
Procedure: Control — Open Debridement alone
  Arms: Control group

SUMMARY:
This study is a prospective, single-center, randomized controlled trial focusing on patients with acute necrotizing pancreatitis (ANP) complicated by pancreatic sinistral portal hypertension (PSPH). The study aims to study the impact of total splenectomy on the debridement efficacy, perioperative recovery, and prognosis of patients with ANP complicated by PSPH.

DETAILED DESCRIPTION:
This study is a prospective, single-center, randomized controlled trial focusing on patients with acute necrotizing pancreatitis (ANP) complicated by pancreatic sinistral portal hypertension (PSPH). A total of 66 participants are planned to be enrolled. The study aims to compare the outcomes of two surgical approaches: open debridement combined with distal pancreatectomy and total splenectomy versus open debridementalone. The objective is to observe the impact of total splenectomy on the debridement efficacy, perioperative recovery, and prognosis of patients with ANP complicated by PSPH. The primary observational indicators include postoperative length of hospital stay, postoperative cost, postoperative life quality, and the alleviation of PSPH. Secondary observational indicators encompass the number of unplanned reoperations, postoperative infection control, postoperative irrigation volume, postoperative antibiotic consumption, and postoperative platelet count change. The study will be carried out in accordance with the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years.
2. Acute necrotic pancreatitis complicated by pancreatic sinistral portal hypertension.
3. Patients undergoing open debridement for infected pancreatic necrosis

Exclusion Criteria:

1. Patients with pre-existing heart, lung, liver, kidney, or other organ failure prior to acute pancreatitis (AP).
2. Patients with pre-existing conditions such as cirrhosis that may lead to portal hypertension prior to AP.
3. Patients with pre-existing hematological diseases prior to AP.
4. Patients undergoing laparoscopic or nephroscopic debridement.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay after debridement | From enrollment of the first subject to completion of follow-up of the last subject (up to 5 years)
  The total length of hospital stay after debridement, including readmissions.
Degree of pancreatic sinistral portal hypertension | From enrollment of the first subject to completion of follow-up of the last subject (up to 5 years)
  The degree of pancreatic sinistral portal hypertension after intervention

SECONDARY OUTCOMES:
Intensive Care Unit stay post Operation | Perioperative
Pancreatic Fistula | Perioperative
  The rate of pancreatic fistula
Number of Draining Tube when Discharged | Perioperative
Time of all draining tubes removal | From enrollment of the first subject to completion of follow-up of the last subject (up to 5 years)
Cost post debridement in the first hospitalization | Perioperative
Number of unplanned re-admissions | From enrollment of the first subject to completion of follow-up of the last subject (up to 5 years)
Number of unplanned operations | From enrollment of the first subject to completion of follow-up of the last subject (up to 5 years)
Number of percutaneous drainage after debridement | From enrollment of the first subject to completion of follow-up of the last subject (up to 5 years)
Antibiotic use after treatment | Perioperative
Abdominal lavage | Perioperative
  Abdominal lavage volume after treatment
Life quality one year after treatment | Within one year after the last subject was treated
  Life quality one year after treatment was judged by the Short-Form 36 Health Survey (SF-36), encompassing both physical and mental health across eight dimensions: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. The minimum value is 0%, the maximum value is 100%, and a higher score means a better life quality.

OTHER OUTCOMES:
Platelet number after debridement | Within one year after the last subject was treated

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No